CLINICAL TRIAL: NCT04520763
Title: Effects of Respiratory Muscle Exercises on Glucose Tolerance in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HOGTT_2020
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Healthy Aging; Healthy Diet

STUDY DESIGN:
Intervention Model Description: This study consists of four visits to the laboratory, each separated by at least 24 hours and each lasting approximately 2.5h. Total duration for each participant is approximately 2 weeks. The study is conducted in 40 healthy adults (≥ 18 years). The study is a randomized, controlled cross-over trial. We chose a cross-over design in order to test the effects of different respiratory exercises compared to a control intervention in order to minimize variability since each subject serves as his/her own control. Due to the nature of the intervention (respiratory muscle exercises), it is not possible to blind participants to the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory Muscle Exercises (Experimental): Two respiratory muscle exercises
  Interventions: Other: 5min respiratory muscle exercises; Other: 15min respiratory muscle exercises
- Control (No Intervention): The control intervention consists of quiet sitting for 15 min

INTERVENTIONS:
Other: 5min respiratory muscle exercises — 5 min of hyperpnea at a target intensity of 60-80% MVV 15-30min after ingestion of 75g of glucose
  Arms: Respiratory Muscle Exercises
Other: 15min respiratory muscle exercises — 5 min of hyperpnea at a target intensity of 60-70% MVV 15-30min after ingestion of 75g of glucose
  Arms: Respiratory Muscle Exercises

SUMMARY:
To evaluate the acute effects of respiratory muscle exercises vs. a control intervention on blood glucose kinetics in healthy adults after an oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Healthy
* Non-smoking
* Body mass index (BMI): 18.5 - 29.9 kg∙m-2
* Normal lung function
* Willing to adhere to study rules

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Intake of medications affecting metabolism, the cardiovascular or the respiratory system, or sleep
* Acute illness or chronic conditions of the gastrointestinal tract, and health conditions affecting metabolism, the cardiovascular or the respiratory system, or sleep
* Pregnancy, breastfeeding, or intention to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Peak blood glucose concentration | throughout the study, an expected average of 2 weeks per participant
  Peak blood glucose concentration will be determined in the three conditions (5min or 15min respiratory muscle exercises or control).
area under the glucose-time curve | throughout the study, an expected average of 2 weeks per participant
  Area under the glucose-time curve will be determined in the three conditions (5min or 15min respiratory muscle exercises or control).

CONTACTS AND LOCATIONS:
Overall Officials: Christin M. Spengler, Prof., Principal Investigator — Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland